CLINICAL TRIAL: NCT06269185
Title: Comparison of Short and Long-term Efficacy Between Infliximab and Adalimumab on Patients With Ulcerative Colitis - a Retrospective Observational Multicenter Cohort Study
Brief Title: Comparison Between Infliximab and Adalimumab on Patients With Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024_IFXvsADAinUC
Record Dates: First submitted 2024-02-09; First posted 2024-02-21 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-03

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: infliximab; adalimumab; anti-TNF therapy
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Infliximab; Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Infliximab: Bio-naive patients with ulcerative colitis who starts treatment with infliximab
  Interventions: Drug: Infliximab
- Adalimumab: Bio-naive patients with ulcerative colitis who starts treatment with adalimumab
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Infliximab — Infliximab is an antiinflammatory drug (anti-TNF therapy) commonly used in treatment of ulcerative colitis
  Groups: Infliximab
Drug: Adalimumab — Adalimumab is an antiinflammatory drug (anti-TNF therapy) commonly used in treatment of ulcerative colitis
  Groups: Adalimumab

SUMMARY:
Anti-TNF (tumor necrosing factor) treatment with infliximab (IFX) and adalimumab (ADA) are established first-line biological therapies used in treatment of patients with ulcerative colitis (UC). There are no head-to-head comparative studies between these two drug but meta-analysis of randomized controlled trials states that IFX might be more effective than ADA for the induction of clinical remission. However, several observational studies conclude that ADA seem to have similar effect as IFX in treating patients with UC but these studies have limitations.

The overall aim of this retrospective multicenter observational cohort study is to evaluate if there is a difference in efficacy between infliximab (IFX) and adalimumab (ADA) in treating bio-naive patients with UC in the short and long term during the modern era when therapeutic drug monitoring have been used to optimize anti-TNF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100 years.
* Diagnosis of ulcerative colitis confirmed by endoscopy and histology.
* Mild, moderate and severe disease activity.
* Initiation of IFX or ADA-treatment at one of the centers of the study.

Exclusion Criteria:

* Clinical remission.
* Previous colonic surgery (resection of colonic segment or colectomy).
* Primary indication for anti-TNF therapy by other disease than UC.
* Prior use of any anti-TNF or other biologic or small molecule therapy.
* Rescue therapy (i.e. infliximab used on hospitalized patients receiving intravenous corticosteroids).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will perform a retrospective multicenter observational cohort study according to the Newcastle-Ottawa Scale (NOS) quality instrument. Bionaive patients (i.e. no prior anti-TNF or other biologic treatment) with active UC, who started treatment with IFX or ADA at four major out-patient IBD-units (Inflammatory Bowel Disease) in the region Västra Götaland in Sweden, will be included in the study. Data regarding exposure for the two compared drugs, baseline characteristics and outcomes after three months and one year will be recieved by a structured review of medical records.
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving steroid-free clinical remission | One year after start of anti-TNF therapy
  Partial Mayo score ≤2 with no subscore >1 and no use of steroids between 6 and 12 months after start of anti-TNF therapy (Partial Mayoscore, range 0-9, with higher value indicating more severe disease activity).

SECONDARY OUTCOMES:
Percentage of patients achieving clinical response | Three months after start of anti-TNF therapy
  A decrease in the partial Mayo score from baseline of 2 or more points, along with either a rectal bleeding subscore of 0 or 1 or a decrease in the rectal bleeding subscore of 1 point or more (Partial Mayoscore, range 0-9, with higher value indicating more severe disease activity).
Percentage of patients achieving clinical remission | Three months after start of anti-TNF therapy
  Partial Mayo score ≤2 with no subscore >1 (Partial Mayoscore, range 0-9, with higher value indicating more severe disease activity).
Percentage of patients achieving biochemical remission | Three months after start of anti-TNF therapy
  Fecal Calprotectin <250 mg/kg
Percentage of patients achieving clinical remission | One year after start of anti-TNF therapy
  Partial Mayo score ≤2 with no subscore >1 (Partial Mayoscore, range 0-9, with higher value indicating more severe disease activity).
Percentage of patients achieving biochemical remission | One year after start of anti-TNF therapy
  Fecal Calprotectin <250 mg/kg
Percentage of patients achieving endoscopic response | 3-12 months after start of anti-TNF therapy
  A decrease in endoscopic Mayo score of 1 or more points (Endoscopic Mayoscore, range 0-3, with higher value indicating more severe disease activity).
Percentage of patients achieving endoscopic remission | 3-12 months after start of anti-TNF therapy
  Endoscopic Mayo score 0-1 (Endoscopic Mayoscore, range 0-3, with higher value indicating more severe disease activity).

OTHER OUTCOMES:
Remission rates in the subpopulations of UC-patients with severe, moderate and mild disease respectively | Three months and one year after start of anti-TNF therapy
  Partial Mayo score ≤2 with no subscore >1 (Partial Mayoscore, range 0-9, with higher value indicating more severe disease activity).

CONTACTS AND LOCATIONS:
Overall Officials: Börje Jonefjäll, PhD, Principal Investigator — Sahlgrenska University Hospital / Mölndal
Locations (1):
- Västra Götalandsregionen, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonovas S, Lytras T, Nikolopoulos G, Peyrin-Biroulet L, Danese S. Systematic review with network meta-analysis: comparative assessment of tofacitinib and biological therapies for moderate-to-severe ulcerative colitis. Aliment Pharmacol Ther. 2018 Feb;47(4):454-465. doi: 10.1111/apt.14449. Epub 2017 Dec 4. PMID 29205421
- [Background] Singh S, Murad MH, Fumery M, Dulai PS, Sandborn WJ. First- and Second-Line Pharmacotherapies for Patients With Moderate to Severely Active Ulcerative Colitis: An Updated Network Meta-Analysis. Clin Gastroenterol Hepatol. 2020 Sep;18(10):2179-2191.e6. doi: 10.1016/j.cgh.2020.01.008. Epub 2020 Jan 13. PMID 31945470
- [Background] Gies N, Kroeker KI, Wong K, Fedorak RN. Treatment of ulcerative colitis with adalimumab or infliximab: long-term follow-up of a single-centre cohort. Aliment Pharmacol Ther. 2010 Aug;32(4):522-8. doi: 10.1111/j.1365-2036.2010.04380.x. Epub 2010 May 25. PMID 20500733
- [Background] Sandborn WJ, Sakuraba A, Wang A, Macaulay D, Reichmann W, Wang S, Chao J, Skup M. Comparison of real-world outcomes of adalimumab and infliximab for patients with ulcerative colitis in the United States. Curr Med Res Opin. 2016 Jul;32(7):1233-41. doi: 10.1185/03007995.2016.1168290. Epub 2016 Mar 30. PMID 26986449
- [Background] Pouillon L, Baumann C, Rousseau H, Choukour M, Andrianjafy C, Danese S, Peyrin-Biroulet L. Treatment Persistence of Infliximab Versus Adalimumab in Ulcerative Colitis: A 16-Year Single-Center Experience. Inflamm Bowel Dis. 2019 Apr 11;25(5):945-954. doi: 10.1093/ibd/izy322. PMID 30329067
- [Background] Lee YI, Park Y, Park SJ, Kim TI, Kim WH, Cheon JH. Comparison of Long-Term Outcomes of Infliximab versus Adalimumab Treatment in Biologic-Naive Patients with Ulcerative Colitis. Gut Liver. 2021 Mar 15;15(2):232-242. doi: 10.5009/gnl19433. PMID 32616683
- [Background] Ma C, Huang V, Fedorak DK, Kroeker KI, Dieleman LA, Halloran BP, Fedorak RN. Outpatient Ulcerative Colitis Primary Anti-TNF Responders Receiving Adalimumab or Infliximab Maintenance Therapy Have Similar Rates of Secondary Loss of Response. J Clin Gastroenterol. 2015 Sep;49(8):675-82. doi: 10.1097/MCG.0000000000000265. PMID 25389599